CLINICAL TRIAL: NCT02767726
Title: A Non-Invasive Cervical Cancer Screening Modality: A Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UPCC 02815
Record Dates: First submitted 2016-05-09; First posted 2016-05-10 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Women With Abnormal Pap Smears

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: non-invasive multimodal imaging

SUMMARY:
Cervix cancer is a major global health concern. A way to screen and immediately treat precancerous lesions (Screen-and-Treat) is greatly needed. Developed by MobileOCT, polarized difference imaging and conventional imaging are used to identify suspicious lesions. We aim to compare this non-invasive method with colposcopy. Patients at the Dickens Clinic will have 3-5 minutes of non-invasive imaging before colposcopy. Pathology will be compared both to colposcopy impression versus MobileOCT.

ELIGIBILITY:
Inclusion Criteria:

* Subjects capable of giving informed consent or have an acceptable surrogate capable of giving consent on subjects behalf.
* Subjects are 18 years of age or older
* Subjects are scheduled for colposcopy clinic based on screening with abnormal pap smear or have repeat colposcopy indicated for specific clinical indications, based off of American Society of Cosposcopy and Cytology.
* Subjects are women.

Exclusion Criteria:

* Pregnancy.
* Males (males do not have a cervix and thus cannot undergo colposcopy).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Number of suspicious lesions identified | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Burkland, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No